CLINICAL TRIAL: NCT01548781
Title: The Effect of Resistance to Participant-Supported Reaching on Workspace of the Hand in Severe Chronic Stroke
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northwestern University (Other)
Collaborators: U.S. Department of Education (U.S. Federal Agency)
Responsible Party: Principal Investigator, Michael Ellis, Assistant Professor, Northwestern University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: H133G110245
Record Dates: First submitted 2012-02-29; First posted 2012-03-08 (Estimated); Last update posted 2015-10-06 (Estimated); Status verified 2015-10

CONDITIONS: Stroke
Keywords: arm; strength; coordination; physical therapy; robotics; stroke; synergy
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Viscous Resistance & Abduction Loading (Experimental): The intervention for the experimental group entails practicing reaching utilizing the robotic device, ACT3D, with the experimental element of horizontal viscosity in combination with abduction loading.
  Interventions: Behavioral: Impairment-based robotic intervention for reaching function
- Abduction Loading (Active Comparator): The intervention for the active comparison group entails practicing reaching utilizing the robotic device, ACT3D, with only abduction loading.
  Interventions: Behavioral: Impairment-based robotic intervention for reaching function

INTERVENTIONS:
Behavioral: Impairment-based robotic intervention for reaching function — All participants will undergo 8 weeks of reaching practice in the ACT3D. Frequency and duration will be matched at three 1.5-hour sessions per week. All reaching practice will include abduction (gravity) loading standardized to the participant's motor abilities. The experimental group intervention will also include a horizontal viscous resistant element similar to pushing the arm through molasses.

SUMMARY:
Disturbances in movement coordination are the least well understood but often the most debilitating with respect to functional recovery following stroke. These deficits in coordination are expressed in the form of abnormal muscle synergies and result in limited and stereotypic movement patterns that are functionally disabling. The result of these constraints in muscle synergies is an abnormal coupling between shoulder abduction and elbow flexion (i.e. the flexion synergy), which significantly reduces the reaching function of an individual with stroke when they lift up the weight of the impaired arm against gravity. The investigators previous neurotherapeutic research, supported by a NIDRR Field Initiated research grant, has shown that the abnormal synergy between shoulder abduction and elbow flexion can be significantly reduced thus increasing total reaching range of motion in individuals with severe stroke. The previous work established progressive abduction loading as a key element to the rehabilitation of reaching. Although individuals with severe stroke benefited from the investigators previous work, residual flexion synergy continued to hinder normal arm function in most participants with severe stroke. This study will utilize the ACT3D robot, developed as part of the investigators previous NIDRR project, to incorporate resistance to reaching while accounting for the known benefits of progressive abduction loading. The investigators propose to randomize forty participants with severe stroke into two closely related interventions. The groups will both practice reaching under abduction loading, however, the experimental group will also move against resistance while reaching. Rigorous and quantitative investigation of therapeutic elements such as resistance to reaching and progressive abduction loading is only possible with a device such as the ACT3D. the investigators will be able to standardize the delivery of each intervention using kinematic and kinetic parameters, which will allow for a clear identification of the therapeutic effect of resistance to reaching. the investigators hypothesize that resistance to reaching in combination with progressive abduction loading will further increase dynamic multi-joint strength, increase total reaching range of motion, and increase arm function thus enhancing actual amount of use of the arm, participation in life roles, and quality of life in individuals with severe stroke.

ELIGIBILITY:
Inclusion Criteria:

* Paresis confined to one side, with substantial motor impairment of the upper limb
* Absence of motor impairment in the unimpaired limb
* Absence of severe concurrent medical problems (e.g. cardiorespiratory impairment, changes in management of hypertension)
* Absence of any acute or chronic painful condition in the upper extremities or spine
* Absence of hemineglect
* Capacity to provide informed consent.

Ages: 21 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2012-03; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
Change in Peak Endpoint Reaching Velocity | Pre-test (Within one week prior to the onset of the intervention) to post-test (Within one week of the final intervention session) & post-test to 3-month follow-up (In the twelfth or thirteenth week following the last intervention session)
  We will quantify peak endpoint reaching velocity with a robotic device, ACT3D, when a participant with stroke reaches as fast as they can toward an outward target under various abduction (gravity) loading conditions. This measure will serve as the primary measure for changes in dynamic multi-joint strength.
Change in Reaching Work Area | Pre-test (Within one week prior to the onset of the intervention) to post-test (Within one week of the final intervention session) & post-test to 3-month follow-up (In the twelfth or thirteenth week following the last intervention session)
  We will quantify total reaching work area (combined shoulder and elbow range of motion) with a robotic device, ACT3D, under various abduction (gravity) loading conditions. This measure will serve as the primary measure changes in dynamic multi-joint range of motion.

SECONDARY OUTCOMES:
Fugl-Meyer Motor Assessment | Pre-(Within one week prior to the onset of the intervention), post-(Within one week of the final intervention session), and 3-month follow up (In the twelfth or thirteenth week following the last intervention session)
  Qualitative and clinical assessment of general motor impairment of arm following stroke.
Rancho Los Amigos Functional Test for the Hemiparetic Upper Extremity | Pre-(Within one week prior to the onset of the intervention), post-(Within one week of the final intervention session), and 3-month follow up (In the twelfth or thirteenth week following the last intervention session)
  Qualitative and clinical assessment of activity limitation (function) of the arm following stroke.
Stroke Impact Scale | Pre-(Within one week prior to the onset of the intervention), post-(Within one week of the final intervention session), and 3-month follow up (In the twelfth or thirteenth week following the last intervention session)
  Structured interview to assess all domains of the ICF (International Classification of Functioning, Disability and Health) in individuals following stroke.
Motor Activity Log | Pre-(Within one week prior to the onset of the intervention), post-(Within one week of the final intervention session), and 3-month follow up (In the twelfth or thirteenth week following the last intervention session)
  Structured interview assessing the individual with stroke's perception of difficulty in the context of arm function during a variety of activities of daily living.

CONTACTS AND LOCATIONS:
Overall Officials: Michael D Ellis, PT, DPT, Principal Investigator — Northwestern University
Locations (1):
- Department of Physical Therapy and Human Movement Sciences, Chicago, Illinois, United States

REFERENCES:
- [Background] Ellis MD, Sukal-Moulton T, Dewald JP. Progressive shoulder abduction loading is a crucial element of arm rehabilitation in chronic stroke. Neurorehabil Neural Repair. 2009 Oct;23(8):862-9. doi: 10.1177/1545968309332927. Epub 2009 May 19. PMID 19454622
- [Background] Ellis MD, Sukal T, DeMott T, Dewald JP. Augmenting clinical evaluation of hemiparetic arm movement with a laboratory-based quantitative measurement of kinematics as a function of limb loading. Neurorehabil Neural Repair. 2008 Jul-Aug;22(4):321-9. doi: 10.1177/1545968307313509. Epub 2008 Mar 8. PMID 18326888
- [Background] Sukal TM, Ellis MD, Dewald JP. Shoulder abduction-induced reductions in reaching work area following hemiparetic stroke: neuroscientific implications. Exp Brain Res. 2007 Nov;183(2):215-23. doi: 10.1007/s00221-007-1029-6. Epub 2007 Jul 20. PMID 17634933
- [Background] Ellis MD, Acosta AM, Yao J, Dewald JP. Position-dependent torque coupling and associated muscle activation in the hemiparetic upper extremity. Exp Brain Res. 2007 Feb;176(4):594-602. doi: 10.1007/s00221-006-0637-x. Epub 2006 Aug 22. PMID 16924488
- [Background] Ellis MD, Holubar BG, Acosta AM, Beer RF, Dewald JP. Modifiability of abnormal isometric elbow and shoulder joint torque coupling after stroke. Muscle Nerve. 2005 Aug;32(2):170-8. doi: 10.1002/mus.20343. PMID 15880629
- [Derived] Ellis MD, Carmona C, Drogos J, Dewald JPA. Progressive Abduction Loading Therapy with Horizontal-Plane Viscous Resistance Targeting Weakness and Flexion Synergy to Treat Upper Limb Function in Chronic Hemiparetic Stroke: A Randomized Clinical Trial. Front Neurol. 2018 Feb 19;9:71. doi: 10.3389/fneur.2018.00071. eCollection 2018. PMID 29515514
- See also: Northwestern University, Feinberg School of Medicine, Department of Physical Therapy and Human Movement Sciences — http://www.feinberg.northwestern.edu/nupthms/